CLINICAL TRIAL: NCT02043236
Title: A Phase II RCT of Strategies to Improve Bone Health in Men on ADT
Brief Title: Strategies to Improve Bone Health in Men on ADT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-6823
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Androgen deprivation therapy; Bone health; Bone mineral density
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy bones pamphlet, letter to GP (Active Comparator): Strategy 1: Written educational material to patient and GP
  Interventions: Behavioral: Healthy bones pamphlet; Behavioral: Letter to GP
- Healthy bones pamphlet, Bone Health Care Coordinator (Active Comparator): Strategy 2: Written educational material to patient and counseling from a Bone Health Care Coordinator
  Interventions: Behavioral: Healthy bones pamphlet; Behavioral: Bone Health Care Coordinator
- Usual care (No Intervention): Control group gets usual care from their oncologist.

INTERVENTIONS:
Behavioral: Healthy bones pamphlet — written educational material
  Other Names: Building strong bones
  Arms: Healthy bones pamphlet, Bone Health Care Coordinator; Healthy bones pamphlet, letter to GP
Behavioral: Bone Health Care Coordinator — The Bone Health Care Coordinator reviews educational materials with participant and facilitates ordering BMD.
  Other Names: BHCC
  Arms: Healthy bones pamphlet, Bone Health Care Coordinator
Behavioral: Letter to GP — The letter to the General Practitioner contains information about the study, recommendations for bone health, guidelines of Osteoporosis Canada, and the identical educational material that the participant received.
  Arms: Healthy bones pamphlet, letter to GP

SUMMARY:
This is a phase II randomized controlled trial (RCT) of 2 strategies to improve bone health in men receiving androgen deprivation therapy (ADT).

DETAILED DESCRIPTION:
In this RCT the investigators are comparing 2 strategies to improve bone health to usual care. Strategy 1 - Patient and physician-specific written educational material. Pilot-tested customized written educational material about bone health for men on ADT will be used for this study. A customized letter will be prepared for the patient's primary care physician, with specific advice and recommendations for the targeted strategies. Both pamphlet and letter will include a list of additional resources. Strategy 2 - patient written material and a bone health care coordinator (BHCC). The same written patient material as in strategy 1 will be used, along with a BHCC who will follow the approach of successful studies and contact the patient by phone or arrange an in-person visit at the hospital if preferred by the patient. The BHCC will also encourage the patient to pursue a bone mineral density test (BMD) with their physician and adopt bone-appropriate diet, lifestyle, and supplement intake recommendations, and will follow up with the patient at least twice over the next 3 months to facilitate behavioural changes and BMD ordering. Counselling sessions are short, typically <15 min. The BHCC will also contact the patient's physician to help facilitate BMD testing. Time points in the study are baseline, 3-month follow up, and 6-month follow up.

Control group The control group consists of a wait-list control for 6 months, during which no specific recommendations or interventions will be made by the study team. Prostate Cancer (PC) clinicians can still provide usual care. At the end of 6 months, control group participants will be referred to the Osteoporosis Clinic at the University Health Network.

ELIGIBILITY:
Inclusion Criteria:

Commencing or planning to continue ADT for a least 6 months 50 years or older English fluency Life expectancy >6 months

Exclusion Criteria:

Prior Bone Mineral Density test within 2 years Prior visit at Osteoporosis Clinic within 2 years

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Patient/physician satisfaction | 6 months
  Satisfaction will be measured with 5-point Likert scale ranging from poor to excellent and administered to patient, PC clinician, and General Physician
Adherence rate | 6 months
  Adherence to following through on recommendations/referrals related to study intervention and clinical outcomes.
Recruitment rate | 6 months
  Enrolled patients divided by approached eligible patients, and reasons for both ineligibility and refusal as documented in logs.
Retention rate | 6 months
  Proportion of patients available for follow-up outcome assessment.
BMD ordering | 6 months
  Rate of Bone Mineral Density ordering

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Alibhai, MD, Principal Investigator — UHN
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alibhai SMH, Breunis H, Timilshina N, Hamidi MS, Cheung AM, Tomlinson GA, Manokumar T, Samadi O, Sandoval J, Durbano S, Warde P, Jones JM. Improving bone health in men with prostate cancer receiving androgen deprivation therapy: Results of a randomized phase 2 trial. Cancer. 2018 Mar 15;124(6):1132-1140. doi: 10.1002/cncr.31171. Epub 2017 Dec 6. PMID 29211305